CLINICAL TRIAL: NCT07301073
Title: The Effect of Postoperative Progressive Relaxation Exercises on Pain, Anxiety, and Physiological Parameters in Emergency General Surgery Patients: A Randomized Controlled Clinical Trial
Brief Title: Postoperative Progressive Relaxation Exercises for Pain and Anxiety After Emergency Surgery
Acronym: PRE-ES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agri Ibrahim Cecen University (Other)
Responsible Party: Principal Investigator, Volkan Gokmen, Asisstant Professor, Agri Ibrahim Cecen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PRE-EMERGENCY-2021
Record Dates: First submitted 2025-11-28; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Emergency Surgical Procedures; Postoperative Pain; Postoperative Anxiety
Keywords: Progressive Relaxation; Emergency Surgery; Postoperative Pain; Anxiety; Physiological Parameters
MeSH Terms: conditions — Pain, Postoperative; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The study used simple computer-generated randomization to allocate participants in a 1:1 ratio to the intervention or control arm. Participants remained in their assigned arm throughout the study.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Outcome assessors who collected pain, anxiety, and physiological measurements were masked to group assignment throughout the study. Data analysts were also blinded by using coded datasets without group identifiers. Participants and care providers could not be masked due to the behavioral nature of the intervention, but standard postoperative care protocols were applied equally to minimize performance bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive Relaxation Exercises (PRE) Intervention (Experimental): Participants assigned to this arm received standardized Progressive Relaxation Exercises (PRE) consisting of three postoperative sessions (each 30 minutes in duration). Sessions were administered at postoperative hour 6, postoperative day 1, and postoperative day 2 by a nurse trained in PRE. The protocol included diaphragmatic breathing, sequential contraction-relaxation of major muscle groups, and a final integration phase. PRE was delivered in addition to routine postoperative care.
  Interventions: Behavioral: Progressive Relaxation Exercises (PRE)
- Routine Postoperative Care Only (No Intervention): Participants in this arm received routine postoperative care according to institutional protocols, including physician-prescribed analgesics, vital sign monitoring, mobilization, wound care, and standard nursing follow-up. No relaxation-based or behavioral intervention was provided. Pain, anxiety, and physiological parameters were assessed at the same scheduled postoperative time points as in the intervention arm.

INTERVENTIONS:
Behavioral: Progressive Relaxation Exercises (PRE) — This intervention consists of structured Progressive Relaxation Exercises (PRE) delivered exclusively in the postoperative period. PRE involves diaphragmatic breathing, awareness of muscle tension, and sequential contraction-relaxation of major muscle groups (hands, arms, shoulders, neck, chest, abdomen, back, hips, legs, and feet). Each session lasts 30 minutes and is administered at the bedside by a nurse trained in PRE. The protocol includes a preparation phase (2-3 min), a muscle relaxation sequence (20-22 min), and an integration phase (3-5 min). PRE is delivered at postoperative hour 6, postoperative day 1, and postoperative day 2, in addition to routine care, and does not include any pharmacological components
  Arms: Progressive Relaxation Exercises (PRE) Intervention

SUMMARY:
This randomized controlled trial investigated the effectiveness of postoperative progressive relaxation exercises (PRE) on pain, anxiety, and physiological parameters among adult patients undergoing emergency general surgery. Seventy patients were randomized to either a PRE intervention delivered at postoperative hour 6, postoperative day 1, and postoperative day 2, or to routine postoperative care. Pain (SF-MPQ), anxiety (STAI), and vital signs were measured. The trial demonstrated that PRE significantly reduced multidimensional pain and anxiety and improved heart rate, respiratory rate, and oxygen saturation. The study provides novel evidence that PRE is feasible and effective when implemented exclusively in the postoperative period among emergency surgical patients.

DETAILED DESCRIPTION:
This randomized, parallel-group clinical trial was conducted to evaluate the effectiveness and feasibility of postoperative progressive relaxation exercises (PRE) among patients undergoing emergency general surgery. Emergency surgical admissions provide no opportunity for preoperative preparation, and postoperative pain, anxiety, and autonomic instability are commonly intensified by acute physiological stress responses. The trial was designed to determine whether PRE, delivered exclusively after surgery, could reduce these symptoms and support early physiological recovery.

Following confirmation of postoperative stability at hour 6, eligible patients were randomly assigned in a 1:1 ratio to either the PRE intervention or routine postoperative care. The intervention consisted of standardized 30-minute sessions of progressive muscle relaxation conducted at postoperative hour 6, postoperative day 1, and postoperative day 2. Sessions followed a structured protocol including diaphragmatic breathing, sequential contraction-relaxation of major muscle groups, and a final integration phase. All sessions were delivered by a nurse trained in PRE.

Outcome assessments were conducted at prespecified time points using validated measures. Pain was evaluated with the Short-Form McGill Pain Questionnaire, anxiety with the State-Trait Anxiety Inventory, and physiological status through routine clinical monitoring of blood pressure, heart rate, respiratory rate, and oxygen saturation. Analyses examined both between-group differences and changes over time.

The study adhered to CONSORT guidelines for randomized trials and incorporated blinded outcome assessment and concealed allocation. No adverse events related to the intervention were reported, and all randomized participants completed follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years or older.
2. Undergoing an emergency surgical procedure requiring postoperative hospitalization.
3. Conscious, oriented, and hemodynamically stable by postoperative hour 6.
4. Able to communicate and follow verbal instructions.
5. No psychiatric, neurological, cognitive, or auditory impairment that would prevent participation.
6. No chronic pain disorder and not using long-term opioids, sedatives, or anxiolytics before admission.
7. Provided written informed consent.

Exclusion Criteria:

1. Postoperative admission to the intensive care unit (ICU).
2. Development of postoperative complications preventing participation (e.g., severe bleeding, respiratory distress, infection).
3. Inability to complete all three scheduled PRE sessions.
4. Postoperative confusion, delirium, or any condition limiting communication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Postoperative Pain Score (SF-MPQ Total Score) | Postoperative hour 6 and postoperative day 2.
  Postoperative pain will be assessed using the Short-Form McGill Pain Questionnaire (SF-MPQ), which includes sensory and affective descriptors, the Present Pain Intensity (PPI) index, and a Visual Analogue Scale (VAS).
  Total Score Range: 0 to 45. Higher scores indicate greater pain severity.
Change in State Anxiety Score (STAI-State, TX-L1) | Postoperative hour 6 and postoperative day 2.
  SSituational anxiety will be assessed using the State Anxiety Inventory (STAI-State).
  Score Range: 20 to 80. Higher scores indicate greater state anxiety.

SECONDARY OUTCOMES:
Change in Trait Anxiety Score (STAI-Trait, TX-L2) | Postoperative hour 6 and postoperative day 2.
  Trait anxiety will be assessed using the STAI-Trait Inventory. Score Range: 20 to 80. Higher scores indicate greater trait anxiety.
Change in Systolic Blood Pressure | Postoperative hour 6, postoperative day 1, postoperative day 2.
  Systolic blood pressure will be measured using a calibrated sphygmomanometer after 10 minutes of rest. Higher values indicate higher systolic blood pressure.
Change in Diastolic Blood Pressure | Postoperative hour 6, postoperative day 1, and postoperative day 2.
  Diastolic blood pressure will be measured using a calibrated sphygmomanometer after 10 minutes of rest.
Change in Heart Rate | Postoperative hour 6, postoperative day 1, and postoperative day 2.
  Heart rate will be measured using bedside monitoring after 10 minutes of rest.
Change in Respiratory Rate | Postoperative hour 6, postoperative day 1, and postoperative day 2.
  Respiratory rate will be measured using standard clinical monitoring after 10 minutes of rest.
Change in Oxygen Saturation (SpO₂) | Postoperative hour 6, postoperative day 1, and postoperative day 2.
  Peripheral oxygen saturation will be measured using pulse oximetry. Higher values indicate better oxygenation.
Use of Nonsteroidal Anti-Inflammatory Drugs (NSAIDs) | Postoperative hour 6, postoperative day 1, and postoperative day 2.
  NSAID use will be recorded at each postoperative assessment based on medication administration records. Higher values indicate greater NSAID consumption.
Use of Opioid Analgesics | Postoperative hour 6, postoperative day 1, and postoperative day 2.
  Opioid analgesic use will be recorded at each postoperative assessment based on medication administration records. Higher values indicate greater opioid consumption.

CONTACTS AND LOCATIONS:
Overall Officials: VOLKAN GÖKMEN, Doctorate, Principal Investigator — Agri ibrahim Cecen Univercity
Locations (1):
- Ağrı Training and Research Hospital, Ağrı, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) from this study will not be shared because the dataset contains sensitive clinical information from emergency surgical patients, and full de-identification cannot be guaranteed without compromising data integrity. Additionally, institutional and national data protection policies restrict the sharing of raw patient-level data outside the hosting institution. Aggregated results and statistical summaries will be made available in publications, but no IPD files will be shared.

REFERENCES:
- [Background] Loh EW, Shih HF, Lin CK, Huang TW. Effect of progressive muscle relaxation on postoperative pain, fatigue, and vital signs in patients with head and neck cancers: A randomized controlled trial. Patient Educ Couns. 2022 Jul;105(7):2151-2157. doi: 10.1016/j.pec.2021.10.034. Epub 2021 Nov 3. PMID 34785078
- [Background] Akinci N. Effect of progressive muscle relaxation on postoperative pain in laparoscopic living kidney donors: a randomized controlled trial. BMC Surg. 2025 Sep 24;25(1):410. doi: 10.1186/s12893-025-03187-y. PMID 40993691
- [Background] Kisaarslan M, Aksoy N. Effect of Progressive Muscle Relaxation Exercise on Postoperative Pain Level in Patients Undergoing Open Renal Surgery: A Nonrandomized Evaluation. J Perianesth Nurs. 2020 Aug;35(4):389-396. doi: 10.1016/j.jopan.2019.12.003. Epub 2020 Mar 24. PMID 32220520
- [Background] Ju W, Ren L, Chen J, Du Y. Efficacy of relaxation therapy as an effective nursing intervention for post-operative pain relief in patients undergoing abdominal surgery: A systematic review and meta-analysis. Exp Ther Med. 2019 Oct;18(4):2909-2916. doi: 10.3892/etm.2019.7915. Epub 2019 Aug 19. PMID 31555379
- [Background] Aslan, F. E. (2006). Ağrı değerlendirilmesi ve ölçümü. In F. E. Aslan (Ed.), Ağrı: Doğası ve Kontrolü (pp. 68-99). İstanbul Tıp Kitabevleri
- [Background] Abbasi, A., Naderi, Z., & Zakerimoghadam, M. (2018). The effect of progressive muscle relaxation on postoperative pain and physiological parameters in patients undergoing abdominal surgery. Journal of PeriAnesthesia Nursing, 33(5), 512-520. https://doi.org/10.1016/j.jopan.2017.11.010